CLINICAL TRIAL: NCT01806714
Title: Text Reminders to Immunize in a Managed Care Organization
Acronym: TRIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Cynthia Rand, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 056103-002
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Human Papilloma Virus
Keywords: HPV vaccination; Adolescent well care; Adolescent HPV immunization; HPV

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text-based reminder for HPV vaccine/WCC (Experimental): Parents of adolescents will receive text-based reminders if their adolescent is due for HPV vaccine (dose 1, 2 or 3) or well child care visit
  Interventions: Other: Text-based reminder for recommended HPV vaccine or WCC
- Control arm (Active Comparator): Parents of adolescents receive preventive health tips via text messages (not specific to services for which child is due)
  Interventions: Other: Non-specific text-based reminder (general health tip)

INTERVENTIONS:
Other: Text-based reminder for recommended HPV vaccine or WCC — Patients due for a well visit or HPV vaccine received a text reminder
  Arms: Text-based reminder for HPV vaccine/WCC
Other: Non-specific text-based reminder (general health tip) — Parents of adolescents receive preventive health tips via text messages (not specific to services for which child is due)
  Arms: Control arm

SUMMARY:
The purpose of the study is to evaluate the effectiveness of a managed care-based HPV vaccination reminder/recall system using a randomized controlled trial (RCT) across diverse practices and patient populations. The trial will measure the effectiveness of text messaging reminder/recall on (a) improving initiation and (b) completion rate of the HPV vaccine series; (c) decreasing the time between vaccine doses; and (d) improving rates of preventive visits for adolescents

The hypotheses are that text-messaged reminders to parents of adolescents will result in improved rates of HPV vaccine series initiation, HPV vaccine series completion, will decrease the intervals between vaccine doses and will improve rates of preventive care among adolescents. Parents receiving specific text-messaged reminders about services (i.e. HPV vaccination, well child care visits) for which their adolescent is due will be compared to a control group of parents receiving general health tips through text messages.

DETAILED DESCRIPTION:
The study setting is western New York State and the Southern Tier of New York State (15 counties total). Investigators will work with the Monroe Plan for Medical Care, an IPA-model managed care organization (MCO) that serves Medicaid managed care and SCHIP enrollees. The MCO will conduct regular reviews of insurance claims data and the New York State Immunization Information System of adolescents ages 11-<16 years. Parents (all over 18 years of age) of adolescents will receive the texted messages on their phones.

There are no enrollment restrictions based upon race or ethnic origin. The inclusion criteria are that the adolescents are a) enrolled in Medicaid or SCHIP through the Monroe Plan, b) have been enrolled greater than 6 months with the Monroe Plan (in order to have sufficient claims data to determine whether they are due for a well child care visit or recommended immunizations), c) the Monroe Plan has received their consent to send preventive care text messages, d) their child attend a primary care practice that has agreed to participate and d) they are between the ages of 11-<16 years at the start of the study.

The key independent measure is group allocation (intervention vs. control); an intention-to-treat strategy will be used to assess the effectiveness of text messaging reminders. Key outcome measures will be: 1) receipt of 0, 1, 2 or 3 doses of HPV vaccine 2) interval (in days) between doses and 3) having a preventive visit in the 6 month period.

ELIGIBILITY:
Inclusion Criteria:

* 11-<18 years
* Member of MCO for >6 months
* Opted in to receive texted reminders from MCO

Exclusion Criteria:

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3812 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Rand, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4182 subjects met eligibility but only a subset were enrolled to receive the intervention because they has functional phone numbers
Pre-assignment Details: For this study, there was a waiver of consent; 4182 subjects met eligibility but only a subset were enrolled to receive the intervention because they has functional phone numbers.
Groups:
- Text-based Reminder for HPV Vaccine/WCC: Parents of adolescents will receive text-based reminders if their adolescent is due for HPV vaccine (dose 1, 2 or 3) or well child care visit
  Text-based reminder for recommended HPV vaccine or well care visit
Period: Overall Study
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm
Started | 2093 | 2089
Completed | 1893 | 1919
Not Completed | 200 | 170
Not completed — No functioning phone number | 200 | 170

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm | Total
Number analyzed (Participants) | 1893 | 1919 | 3812
Age, Customized [Number; unit: participants]
  11 year olds | 428 | 407 | 835
  12 year olds | 341 | 380 | 721
  13 year olds | 307 | 324 | 631
  14 year olds | 281 | 288 | 569
  15 year olds | 271 | 270 | 541
  16 year olds | 265 | 250 | 515
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 863 | 868 | 1731
  Male | 1030 | 1051 | 2081

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Receiving HPV Vaccination (Dose 1)
Description: Participants who received HPV vaccine dose 1 Kaplan-Meier failure function
Time Frame: 9 months
Population: Only subjects with valid phone numbers at the time dose 1 was dispensed received dose 1.
Measure: Number; unit: percentage of eligible participants
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm
Number analyzed (Participants) | 964 | 961
percentage of eligible participants | 16 | 13
Statistical Analysis 1: Comparison: Text-based Reminder for HPV Vaccine/WCC vs Control Arm; Test type: Superiority or Other; p < 0.04, clustered stratified Proportional Hazard; Cox Proportional Hazard = 1.3, 95% CI 2-sided [1.0 to 1.6] — We determined hazard ratios using a clustered stratified Cox model with the Efron method to handle tied events and the Huber/White variance estimator that clustered on primary care provider and stratified on practice

2. Secondary Outcome: Percentage of Participants Receiving HPV Vaccination (Dose 2)
Description: Participants who received HPV vaccine dose 2 at end of study period Kaplan-Meier failure function
Time Frame: 9 months
Population: Only subjects with a valid phone number at the time dose 2 was dispensed received the vaccine. The number of subjects receiving dose 2 is higher than dose 1 because some phones numbers that were inactive during dose 1 were active during dose 2.
Measure: Number; unit: percentage of eligible participants
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm
Number analyzed (Participants) | 1007 | 1014
percentage of eligible participants | 6 | 7

3. Secondary Outcome: Percentage of Participants Receiving HPV Vaccination (Dose 3)
Description: Participants who received HPV vaccine dose 3 at end of study period Kaplan-Meier failure function
Time Frame: 9 months
Population: Only subjects with valid phone numbers were included and not all recipients got the 2nd dose. Only subjects who got the 2nd dose were then given the 3rd dose and only if they had working phone numbers.
Measure: Number; unit: percentage of eligible participants
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm
Number analyzed (Participants) | 958 | 966
percentage of eligible participants | 2 | 2

ADVERSE EVENTS:
Time Frame: July 2013 - December 2014
Arm/Group | Text-based Reminder for HPV Vaccine/WCC | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/1893 | 0/1919
Other Adverse Events (participants affected / at risk) | 0/1893 | 0/1919

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No